CLINICAL TRIAL: NCT06121622
Title: Development of New Personalised 3D Preclinical Models of Pancreatic Neuroendocrine Tumours
Acronym: 3DPanNET
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Anna Battistella, Principal Investigator, IRCCS San Raffaele
Other Study IDs: 3DPanNET
Record Dates: First submitted 2023-10-26; First posted 2023-11-08 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Neuroendocrine Tumor
Keywords: PanNET; 3D preclinical models
MeSH Terms: conditions — Adenoma, Islet Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour surgical samples not required for diagnostic procedures, will be employed for the generation of personalised 3D preclinical models
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this prospective observational study is to generate new personalised 3D preclinical models of pancreatic neuroendocrine tumors. The models will be exploited for studying the mechanisms underlying disease development and progression, as well as for performing drug testing. For the development of the newly proposed models, patients' surgical specimens will be evaluated by the Pathological Unit. If the presence of pathological material in excess, not required for the routine diagnostic procedure, is confirmed, such material will be employed for the generation of the proposed personalised models.

DETAILED DESCRIPTION:
Pancreatic neuroendocrine tumors (PanNETs) are characterized by highly heterogeneous biological behavior. Another distinctive feature of these neoplasms is the presence of a dense vascular network, reminiscent of their physiological counterpart. Indeed, the tumor microenvironment plays a critical role in these neoplasms and influence their therapeutic management. Although they are typically indolent in nature, approximately 40% of PanNET patients are metastatic at diagnosis, requiring non-surgical treatments such as somatostatin therapy, chemotherapy, targeted therapy, and peptide receptor radionuclide therapy (PRRT). Furthermore, 1 out of 5 patients experience disease recurrence after surgical resection, necessitating pharmacological therapies. Currently, no specific recommendations exist on the most effective therapeutic sequence to follow in presence of metastatic disease/disease relapse. One of the main reasons behind this unmet clinical need is the scarcity of available preclinical models of these neoplasms able to accurately reproduce the biology and physiology of the primary tumor and that can be used as valid platforms for drug testing.

The study aims to generate a new 3D in vitro model of PanNET, replicating the complex primary tumor in vitro, including also the tumor microenvironment (e.g., vascular network and stroma, essential elements of these neoplasms), personalised for each patient. Indeed, for the development of the newly proposed models, patients' surgical specimens will be initially evaluated by the Pathological Unit and, in the presence of pathological material in excess not required for the routine diagnostic procedure, it will be employed for the generation of the proposed personalised models. 3D culture techniques (e.g., 3D bioprinting) will be used for the development of the models. Moreover, in order to further mimic in vitro the in vivo environment, the models will be maintained under dynamic conditions.

These newly proposed models will be exploited for studying the mechanisms underlying disease development and progression, as well as for performing drug testing.

ELIGIBILITY:
Inclusion criteria:

* patients who undergo pancreatic surgical resection for non-functioning pancreatic neuroendocrine tumor
* age ≥ 18 years
* informed consent

Exclusion criteria:

* non-pancreatic neuroendocrine tumor histological diagnosis
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total number of approximately 70 patients will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Development of New Personalised 3D Preclinical Models of Pancreatic Neuroendocrine Tumours | from the day of surgery until 3 years from surgery
  Generation of new 3D preclinical models of pancreatic neuroendocrine tumors for the study of the disease biology and for the assessment of drug response

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffele Institute, Milan, MI, Italy